CLINICAL TRIAL: NCT02168543
Title: Clinical Efficacy of Subgingivally Delivered 1% Alendronate in the Treatment of Smokers With Chronic Periodontitis: a Randomized Placebo Controlled Clinical Trial.
Brief Title: 1% Alendronate Gel in Treatment of Chronic Periodontitis Among Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. Anuj Sharma, Anuj Sharma, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GDCRI-09-03
Record Dates: First submitted 2014-06-11; First posted 2014-06-20 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Alendronate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alendronate (Experimental): 1% Alendronate gel once in periodontal pocket (Gums)
  Interventions: Drug: Alendronate
- Placebo (Placebo Comparator): Placebo gel once in periodontal pocket (Gums)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alendronate
  Arms: Alendronate
Drug: Placebo
  Arms: Placebo

SUMMARY:
* Locally delivered Alendronate (ALN) have potent inhibitory effect on bone and increases new bone formation in chronic periodontitis patients
* Till date no study has reported the effect of local delivery of ALN in chronic periodontitis patients among smokers. Hence the aim of this study is to investigate the clinical and radiographic effects of locally delivered ALN as an adjunct to the non surgical treatment in smoker chronic periodontitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy subjects with probing depth (PD) ≥ 5 mm or periodontal attachment level (PAL) ≥ 4 to 6 mm and a radiographical vertical bone loss ≥ 3 mm
* No history of periodontal therapy in preceding last 6 months
* No use of antibiotics in the preceding 6 months

Exclusion Criteria:

* Subjects with known systemic disease
* Known or suspected allergy to the ALN/bisphosphonate group
* Those on systemic ALN/bisphosphonate therapy
* Subjects with aggressive periodontitis,
* Use of smokeless tobacco in any form,
* Alcoholics
* Immunocompromised subjects
* Pregnant or lactating females

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2009-03; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline plaque scores at 2 month and 6 month | At baseline, 2nd month and 6th month
  Plaque scores assessed at baseline, at 2 months and 6 months for Alendronate and placebo group
Change from baseline gingival scores at 2 month and 6 month | At baseline, 2nd month and 6th month
  Gingival scores assessed at baseline, at 2 months and 6 months for Alendronate and placebo group

SECONDARY OUTCOMES:
Change from baseline Probing depth at 2 month and 6 month | At baseline, 2nd month and 6th month
  Probing depth assessed at baseline, at 2 months and 6 months for Alendronate and placebo group
Change from baseline Periodontal attachment level at 2 month and 6 month | At baseline, 2nd month and 6th month
  Periodontal attachment level assessed at baseline, at 2 months and 6 months for Alendronate and placebo group
Change from baseline intrabony defect depth at 6 month | At baseline and 6th month
  intrabony defect depth assessed at baseline and 6 months for Alendronate and placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anuj Sharma, BDS, MDS, Principal Investigator — RIMS, Ranchi